CLINICAL TRIAL: NCT02824965
Title: A Phase I/II Open-label Trial of Intravenous CAVATAK^TM in Combination With Pembrolizumab for the Treatment of Patients With Advanced NSCLC
Brief Title: Pembrolizumab + CVA21 in Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2015-001
Record Dates: First submitted 2016-06-13; First posted 2016-07-07 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+1x10^9 TCID50 CVA21 (Experimental): CVA21 will be administered IV on days: 1, 3, 5, 8 29, 50, 71, 92, 113 134, and 155. 200mg Pembrolizumab will be administered as per normal dosing frequency at Q3W IV, and will continue for up to 24 months. Should dose limiting toxicities be observed participants may be transferred a lower dosage of CVA21.
  Interventions: Drug: Pembrolizumab; Biological: CVA21

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a selective monoclonal antibody that blocks the interaction between PD1 and its ligands PDL1 and PDL2, resulting in infiltration of tumour specific CD8+ T-cells and ultimately leads to tumour rejection.
  Other Names: KEYTRUDA
Biological: CVA21 — CAVATAK is an oncolytic Coxsackie virus that specifically infects and kills ICAM overexpressing tumour cells
  Other Names: CAVATAK, Coxsackie virus 21

SUMMARY:
This will be a Phase Ib open-label trial of CAVATAK™ (CVA21) in combination with Pembrolizumab for the treatment of patients with advanced NSCLC. The dose of Pembrolizumab will be fixed at 200mg. Three cohorts (dose levels) of intravenously-delivered CVA21 will be explored, using a standard 3+3 patient dose escalation design. The starting dose of CVA21 will be one log below the 1 x 10^9 TCID50 dose found to be safe when CVA21 was given alone in an ongoing Phase I study (NCT02043665).

DETAILED DESCRIPTION:
Primary Objective & Hypothesis

(1) Objective:

To evaluate the safety of intravenous CVA21 in combination with pembrolizumab in patients with advanced NSCLC.

Hypothesis:

Pembrolizumab in combination with intravenous CVA21 will be well tolerated in patients with advanced NSCLC.

Secondary Objective & Hypothesis

(1) Objective:

i. To evaluate the efficacy of intravenous CVA21 in inducing an immune cell rich tumour microenvironment in patients with a baseline biopsy demonstrating a tumour with an immune cell poor microenvironment.

ii. To evaluate the efficacy of intravenous CVA21 in combination with pembrolizumab in patients with advanced NSCLC using irRECIST.

iii. To evaluate the safety of intravenous CVA21 in combination with pembrolizumab.

iv. To identify a safe and potentially effective dose for intravenous CVA21 in combination with intravenous pembrolizumab.

v. To serially evaluate the presence of detectable virus and anti-viral antibodies in peripheral blood of the trial participants.

Hypothesis:

i. CVA21 will induce immune cell infiltration into tumors of patients that lack an immune cell rich micro-environment.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
5. Have a performance status of 0 - 1 on the ECOG Performance Scale.
6. Histologically confirmed NSCLC.
7. No CVA21 neutralising antibody (≤ 1:16).
8. Life expectancy > 3 months.
9. Acceptable haematological, renal and hepatic function.
10. Protocol approved by local Research Ethics Committees.
11. No chemotherapy, radiation therapy, hormonal treatment of immunotherapy within 28 days of dosing, except small doses of RT (<20 Gy) given for symptomatic bone metastases.
12. Have resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia). If subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
13. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in section 6.13.2, starting with the first dose of study drug therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. Male subjects of child-bearing potential must agree to use an adequate method of contraception outlined in section 6.13.2, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
16. Failed at least one line of standard chemotherapy or tyrosine kinase inhibitor (TKI) as treatment for Stage IV NSCLC. Patients with EGFR mutations or ALK gene rearrangements are eligible only after initial TKI failure and chemotherapy is not felt to be a suitable option by the investigator.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has active cardiac disease.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has a history of interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has previously received treatment with CVA21.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | 0-24 months
  To evaluate the safety of intravenous CVA21 in combination with pembrolizumab in patients with advanced NSCLC. All adverse events will be collected and assessed with regards to CTCAE V4.0 grading, seriousness, duration and relationship to the study drugs.

SECONDARY OUTCOMES:
ORR from the date of first study treatment as assessed by RECIST | 0-24 months
  Quantification of the Objective Response rate in patients on study by RECIST
ORR from the date of first study treatment as assessed by immune related response criteria (irRC) | 0-24 Months
  The overall response according to the irRC is derived from time-point response assessments based on tumor burden. In the irRC, an immune-related Complete Response (irCR) is the disappearance of all lesions, measured or unmeasured, and no new lesions; an immune-related Partial Response (irPR) is a 50% drop in tumour burden from baseline as defined by the irRC; and immune-related Progressive Disease (irPD) is a 25% increase in tumour burden from the lowest level recorded. Everything else is considered immune-related Stable Disease (irSD).
PFS | 0-36 Months
  Progression Free survival from first study treatment until end of study
Incidence of detectable CVA21 virus and neutralizing antibodies | 0-24 Months
  Measurement of CVA21 virus and neutralizing antibodies at each CVA21 injection time point
OS | 0-36 Months
  Overall survival of patients on study from first study treatment.
Change in PD-L1 expression from sequential biopsies in NSCLC patients | 0-36 months
  PD-L1 expression will be measured using IHC from baseline and sequential biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Thomas John, Principal Investigator — Austin Health
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No